CLINICAL TRIAL: NCT01334515
Title: Feasibility/Phase II Study of hu14.18-IL2 Immunocytokine + GM-CSF and Isotretinoin in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Biological Therapy, Sargramostim, and Isotretinoin in Treating Patients With Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL1021; NCI-2011-02672 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000698589 (Other: Clinical Trials.gov); U10CA098543 (NIH); COG-ANBL1021 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lorukafusp alfa; Isotretinoin; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disease measured by standard radiographic criteria (Experimental): Treatment (hu14.18-Interleukin 2(IL2) fusion protein and isotretinoin). Patients receive sargramostim (SC [preferred]) or IV over 2 hours on days 1-2 and 8-14, hu14.18-IL2 fusion protein IV over 4 hours on days 4-6, and isotretinoin PO twice daily on days 11-24. Treatment repeats every 28 days for 4-10 courses in the absence of disease progression or unacceptable toxicity. Patients in stratum-1 who achieve stable disease (SD) after course 4 are removed from protocol therapy. Patients in stratum-2 who achieve SD after course 4 receive 2 additional courses of study treatment. Patients may undergo blood and bone marrow sample collection periodically for correlative studies.
  Interventions: Biological: hu14.18-IL2 fusion protein; Drug: isotretinoin; Biological: sargramostim; Other: laboratory biomarker analysis
- Disease evaluable only by I-MIBG or BM histology (Experimental): Treatment (hu14.18-Interleukin 2(IL2) fusion protein and isotretinoin). Patients receive sargramostim (SC [preferred]) or IV over 2 hours on days 1-2 and 8-14, hu14.18-IL2 fusion protein IV over 4 hours on days 4-6, and isotretinoin PO twice daily on days 11-24. Treatment repeats every 28 days for 4-10 courses in the absence of disease progression or unacceptable toxicity. Patients in stratum-1 who achieve stable disease (SD) after course 4 are removed from protocol therapy. Patients in stratum-2 who achieve SD after course 4 receive 2 additional courses of study treatment. Patients may undergo blood and bone marrow sample collection periodically for correlative studies.
  Interventions: Biological: hu14.18-IL2 fusion protein; Drug: isotretinoin; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: hu14.18-IL2 fusion protein — Given IV
  Other Names: EMD 273063; hu14.18-IL2
Drug: isotretinoin — Given PO
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well hu14.18-interleukin-2 (IL2) fusion protein works when given together with sargramostim and isotretinoin in treating patients with relapsed or refractory neuroblastoma. Biological therapy, such as hu14.18-IL2 fusion protein, and sargramostim work in different ways to stimulate the immune system and stop tumor cells from growing. Drugs used in chemotherapy, such as isotretinoin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving hu14.18-IL2 fusion protein together with sargramostim and isotretinoin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of sargramostim (GM-CSF) and isotretinoin given in combination with hu14.18-IL-2 (hu14.18-IL2 fusion protein), as a test of feasibility for a future Phase III study.

II. To evaluate the anti-tumor activity of hu14.18-IL2 given in combination with GM-CSF and isotretinoin in patients with recurrent or refractory neuroblastoma with disease measurable by standard radiographic criteria (stratum-1).

III. To evaluate the anti-tumor activity of hu14.18-IL2 given in combination with GM-CSF and isotretinoin in patients with recurrent or refractory neuroblastoma evaluable only by meta iodo benzyl guanidine I 123 (MIBG) scintigraphy and/or bone marrow histology (stratum-2).

SECONDARY OBJECTIVES:

I. To describe the disease burden of stratum-2 patients by semi-quantitative assessment of bone marrow and MIBG scintigraphy and determine whether there is an association between lower disease burden and response to hu14.18-IL2.

II. To assess molecular parameters of response (reverse-transcriptase (RT) polymerase chain reaction (PCR)) for patients meeting complete response (CR) criteria.

III. To evaluate the immunologic activation induced in vivo by hu14.18-IL2. IV. To determine the induction of anti-hu14.18-IL2 antibody by treatment with hu14.18-IL2.

V. To test for associations between tumor response versus immune activation and anti-hu14.18-IL2 activity, and between measurements of toxicity versus immune activation and anti-hu14.18-IL2 activity.

OUTLINE: This is a multicenter study. Patients are stratified according to measurable disease (disease measurable by standard radiographic criteria [stratum-1] vs disease evaluable only by meta iodo benzyl guanidine I 123 (MIBG) and/or bone marrow histology [stratum-2]).

Patients receive sargramostim subcutaneously (SC [preferred]) or IV over 2 hours on days 1-2 and 8-14, hu14.18-IL2 fusion protein IV over 4 hours on days 4-6, and isotretinoin orally (PO) twice daily on days 11-24. Treatment repeats every 28 days for 4-10 courses in the absence of disease progression or unacceptable toxicity. Patients in stratum-1 who achieve stable disease (SD) after course 4 are removed from protocol therapy. Patients in stratum-2 who achieve SD after course 4 receive 2 additional courses of study treatment. Patients may undergo blood and bone marrow sample collection periodically for correlative studies.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 2 years, and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* The target tumor is limited to neuroblastoma; patients must have had histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines at the time of initial diagnosis
* Patients must have resistant/refractory or recurrent neuroblastoma
* Tumor imaging and bone marrow evaluation for histologic analysis of marrow tumor cell quantity must be obtained within 3 weeks (21 days) prior to enrollment onto study and patients must have one of the following:

  * Measurable tumor on magnetic resonance imaging (MRI), computed tomography (CT) scan, or x-ray defined as minimum of 20 mm in at least one dimension; measurable is defined as minimum of 20 mm in at least one dimension; for patients who are in first response (i.e., those patients with persistent sites of tumor after frontline therapy, but who have never relapsed), a biopsy of a lesion or bone marrow must demonstrate viable neuroblastoma following completion of therapy; if the lesion was irradiated, the biopsy must be done at least 4 weeks after radiation is completed
  * Meta iodo benzyl guanidine I 123 (MIBG) scan with positive uptake at minimum of one site; for patients in first response, a biopsy of site must demonstrate viable tumor; if lesion was radiated, biopsy must be done at least 4 weeks after radiation completed
  * Bone marrow with tumor cells seen on routine morphology (not by neuron specific enolase (NSE) staining only) of bilateral aspirate and/or biopsy on one bone marrow sample
* Patients must have a performance status of 0, 1 or 2; use Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age
* Patients must have a life expectancy of ≥ 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Myelosuppressive chemotherapy: Must not have received within 3 weeks of entry onto this study (4 weeks if prior nitrosourea).
* Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a non-myelosuppressive biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; for information on half-lives of these agents, refer to the table provided in the following link: https://members.childrensoncologygroup.org/_files/disc/dvl/Half-lifetableforeligibility.pdf
* External beam radiation therapy (XRT): >= 2 wks for local palliative XRT (small port); >= 6 months must have elapsed if prior craniospinal XRT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* Autologous stem cell transplant (ASCT): Patients are eligible > 56 days after autologous stem cell infusion following myeloablative therapy; patients receiving an autologous stem cell infusion to support non-myeloablative therapy (including 131I-MIBG given as a single agent) are eligible at any time as long as they meet the hematologic and other organ function criteria for eligibility; patients who have received an allogenic stem cell transplant are excluded
* radioactive iodine (131 I) MIBG therapy: Patients are eligible > 6 weeks after therapeutic 131I-MIBG
* Study specific limitations on prior therapy: Subjects who have previously received in vivo anti-GD2 monoclonal antibodies for biologic therapy or for tumor imaging, are eligible unless they have had progressive disease or a severe allergic reaction while receiving prior anti-disialoganglioside (GD2) therapy; subjects who have received autologous marrow infusions or autologous stem cell infusions using monoclonal antibody linked to beads to purge specimens, but no other form of anti-GD2 monoclonal antibody, are eligible
* Growth factor(s): Must not have received within 1 week of entry onto this study
* Steroids: Patients who require or are likely to require corticosteroid or other immunosuppressive drugs for intercurrent disease (any other significant medical problem related to or independent from the neuroblastoma or its treatment) while tentatively scheduled to be receiving treatment on this study are ineligible; the only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product transfusion in order to avoid allergic transfusion reactions
* Peripheral absolute phagocyte count (APC=neutrophils + monocytes) >= 1000/uL
* Platelet count ≥ 20,000/μL*
* Hemoglobin ≥ 8 g/dL*
* Transfusions are permitted to meet these platelet and hemoglobin criteria, if the patient is known to have a history of bone marrow involvement with tumor; patients with platelet counts < 20,000/uL who are refractory to platelet transfusions are not eligible for this study; patients requiring transfusions of platelets or red blood cells (RBC) to meet eligibility criteria will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min OR serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 years of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5 x upper limit of normal (ULN) for age
* Shortening fraction of >= 27% by echocardiogram
* Ejection fraction of >= 55% by gated radionuclide study (interleukin 2 [IL2] is associated with capillary leak and, at high doses, pulmonary edema)
* Corrected QT (QTC) interval < 450 msec
* Due to risk of IL2 associated vascular leak and pulmonary edema, patients must have normal respiratory function; this is defined as no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% on room air; if pulmonary function tests (PFTs) are performed, the forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) must be greater than 60%
* Patients with a history of central nervous system (CNS) disease must have no clinical or radiological evidence of CNS disease at the time of protocol enrollment; (it is currently unknown whether hu14.18-IL2 penetrates the blood brain barrier to provide effective CNS treatment)
* Patients with seizure disorders may be enrolled if on anti-convulsants and well-controlled
* CNS toxicity =< grade 2

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test
* Patients of childbearing potential must agree to use an effective birth control method (as isotretinoin is known to be teratogenic)
* Female patients who are lactating must agree to stop breast-feeding
* Patients with symptoms of congestive heart failure or uncontrolled cardiac rhythm disturbance are not eligible
* Patients with symptomatic pleural effusions or ascites (requiring constant or intermittent drainage) because IL2 is associated with capillary leak are not eligible
* Patients who have had major surgery (i.e., laparotomy or thoracotomy) within the past 2 weeks are not eligible, due to the capillary leak associated with IL2
* Patients with organ allografts (including bone marrow or stem cell) due to the immune activating effects of IL2 are not eligible; patients receiving prior autologous bone marrow or stem cell re-infusions are eligible
* Patients with prior history of ventilator support related to lung injury (lung injury such as pneumonia, hemorrhagic pneumonitis, capillary leakage) are excluded
* Patients with significant serious intercurrent illnesses (any other ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and which is expected to interfere with the action of hu14.18-IL2 or to significantly increase the severity of the toxicities experienced from hu14.18-IL2 treatment are not eligible

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12-31 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Shusterman, MD, Principal Investigator — Children's Oncology Group
Locations (76):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Oncology Group, Arcadia, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Childrens Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Raymond Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie W Bryant Cancer Center, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Hospital Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Disease Measured by Standard Radiographic Criteria; Disease Evaluable Only by I-MIBG or BM Histology: Treatment (hu14.18-IL2 fusion protein and isotretinoin). Patients receive sargramostim (SC [preferred]) or IV over 2 hours on days 1-2 and 8-14, hu14.18-IL2 fusion protein IV over 4 hours on days 4-6, and isotretinoin PO twice daily on days 11-24. Treatment repeats every 28 days for 4-10 courses in the absence of disease progression or unacceptable toxicity. Patients in stratum-1 who achieve SD after course 4 are removed from protocol therapy. Patients in stratum-2 who achieve SD after course 4 receive 2 additional courses of study treatment. Patients may undergo blood and bone marrow sample collection periodically for correlative studies.
  hu14.18-IL2 fusion protein: Given IV
  isotretinoin: Given PO
  sargramostim: Given SC
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Disease Measured by Standard Radiographic Criteria | Disease Evaluable Only by I-MIBG or BM Histology
Started | 16 | 36
Completed | 4 | 7
Not Completed | 12 | 29
Not completed — Adverse Event | 1 | 6
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 8 | 21
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disease Measured by Standard Radiographic Criteria | Disease Evaluable Only by I-MIBG or BM Histology | Total
Number analyzed (Participants) | 16 | 36 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.94 [4.30 to 9.80] | 8.75 [5.79 to 12.38] | 8.31 [5.39 to 11.37]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 32 | 47
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 10 | 24 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 25 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 11 | 30 | 41
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 33 | 47
  Canada | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Unacceptable Dose Limiting Toxicities (DLTs)
Description: Test for tolerability and monitor for the occurrence of too many unacceptable DLTs using a two-stage stopping rule: (Stage 1) Accrue 10 patients. If more than 1 experience at least one unacceptable DLT during the first treatment cycle, the regimen will be considered to have unacceptable toxicity, and accrual will be temporarily closed, to review all relevant data and consider modifying the regimen to improve safety. If 1 or no patients have an unacceptable DLT in the first treatment cycle, then continue. (Stage 2) Accrue 20 more patients. If 7 or more experience at least one unacceptable DLT in the first treatment cycle, temporarily close the study for possible dosing-safety modifications. If 6 or fewer have an unacceptable DLT in the first treatment cycle, it is reasonable to assume that the combination therapy is safe.
Time Frame: Up to 10 courses
Population: This outcome measure evaluates the first 30 patients to enroll and who receive at least one dose of hu14.18-IL2.
Measure: Number; unit: participants
Arm/Group | Disease Measured by Standard Radiographic Criteria | Disease Evaluable Only by I-MIBG or BM Histology
Number analyzed (Participants) | 10 | 20
participants
  Patients with Unacceptable DLTs | 1 | 2
  Patients without Unacceptable DLTs | 9 | 18

2. Secondary Outcome: Overall Response Evaluated in This Study Using the New International Criteria Proposed by the Revised Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of patients where best overall response is a complete response (CR)-[disappearance of all target lesions and disappearance of any other measureable disease], a very Good Partial Response (VGPR)- [>90% decrease of the disease measurement for CT/MRI lesions, taking as reference the disease measurement done to confirm measurable disease at study entry. Non-target CT/MRI lesions stable to smaller in size], or partial Response (PR)- [>= 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study entry. Non-target CT/MRI lesions stable to smaller in size], and maintains the response. It is possible that a subject's response to therapy may not occur until after several months of treatment. In order to prevent bias, the maximum duration of time/treatment over which a subject's response is to be assessed for determination of the best overall response is after the completion of up to 10 courses.
Time Frame: Every two cycles (each cycle lasts 28 days)
Population: Patients will be evaluable for inclusion in the analysis of response if they have an event at any time on the study or if they complete at least 2 cycles of hu14.18-IL2 therapy. Patients who go off-protocol therapy prior to the completion of 2 cycles due to parent/family choice and/or due to toxicity will not be considered evaluable for response.
Measure: Number; unit: participants
Arm/Group | Disease Measured by Standard Radiographic Criteria | Disease Evaluable Only by I-MIBG or BM Histology
Number analyzed (Participants) | 15 | 30
participants
  Responders | 1 | 6
  Non-Responders | 14 | 24

ADVERSE EVENTS:
Description: SAE field contains NCI Common Toxicity Criteria for Adverse Effects (CTCAE) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Only Grade 3 and higher Adverse Events were collected/assessed in this study.
Arm/Group | Disease Measured by Standard Radiographic Criteria | Disease Evaluable Only by I-MIBG or BM Histology
Serious Adverse Events (participants affected / at risk) | 7/16 | 18/36
Other Adverse Events (participants affected / at risk) | 13/16 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Measured by Standard Radiographic Criteria (N=16) | Disease Evaluable Only by I-MIBG or BM Histology (N=36)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 4 (5) | 6 (7)
GGT increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 3 (4) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Measured by Standard Radiographic Criteria (N=16) | Disease Evaluable Only by I-MIBG or BM Histology (N=36)
Anemia (Blood and lymphatic system disorders) | 9 (11) | 11 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 10 (22)
Pain (General disorders) | 2 (2) | 6 (10)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 2 (4) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 14 (20)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 11 (13)
Blood bilirubin increased (Investigations) | 2 (4) | 4 (10)
GGT increased (Investigations) | 0 (0) | 2 (4)
Lymphocyte count decreased (Investigations) | 2 (3) | 10 (16)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (6)
Platelet count decreased (Investigations) | 5 (7) | 11 (20)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (2) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 3 (6)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.